CLINICAL TRIAL: NCT03845816
Title: L'évaluation de l'Attachement, de l'Auto-compassion et Des stratégies de Coping Chez Les Patients Douloureux Chroniques
Brief Title: Evaluation of Attachment, Self-compassion and Coping Strategies in Chronic Pain Patients
Acronym: attachpain
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-A01167-48
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Self-Compassion Scale (SCS) questionnaire — all included patients with chronic pain will answer the Self-Compassion Scale (SCS) questionnaire

SUMMARY:
Compare the self-compassionate score by type of attachment, "safe" or "insecure", in chronic pain patients.

DETAILED DESCRIPTION:
Attachment theory proposes a theoretical model that helps us explain how the process of developing interpersonal relationships can affect the search for care and the response of individuals to an illness.

Self-compassion is a concept developed by Kristin Neff. It refers to the disposition of each individual to contain their feelings of suffering by a feeling of warmth, connection and care.

The coping corresponds to the answers, the reactions, that the individual will develop to control, reduce or simply tolerate the aversive situation. Coping can take the form of cognitions, affects and behaviors that an individual will put in place to deal with a situation.

The three concepts (attachment, self-compassion, coping) seem to be interrelated, and they contribute to the explanation and management of chronic pain, in the spectrum of the bio-psycho-social model of pain. Yet no study has measured these three variables together in chronic pain patients

Chronic and Newly Assisted Patients at CETD (Neurosurgery Department, Pain Assessment and Treatment Center) (ie any patient seen for the first time in pain center, and included in the research during one of the three medical consultations preliminary to overall care at the CETD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain

Exclusion Criteria:

* Legal protection measure
* Patients followed for cancer
* Patients followed for multiple sclerosis
* Patients followed for Parkinson's disease
* Patients already followed in another CETD
* Decompensated psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient newly treated at the pain center (i.e. any patient seen for the first time in a pain centre, and included in the research during one of the three medical consultations preliminary to overall management at the patient center)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Quetionnaire | 1 month
  The self-compassion score level according to the Self-Compassion Scale Questionnaire (SCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided